CLINICAL TRIAL: NCT01360424
Title: Efficacy of Teriparatide Treatment in Patients With New Forms of Inherited Low-Turnover Osteoporosis
Brief Title: Teriparatide Treatment in Patients With Inherited Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Ville-Valtteri Välimäki, Dr, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS-LTO-PTH; 2010-019297-32 (EudraCT Number)
Record Dates: First submitted 2011-05-06; First posted 2011-05-25 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis
Keywords: osteoporosis; teriparatide; bone turnover; New forms of inherited low-turnover osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- teriparatide (Experimental)
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Daily administration of teriparatide 20 ug s.c. for 24 months

SUMMARY:
The purpose of this study is to analyse efficacy of teriparatide treatment in patients with new forms of inherited low-turnover osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* inherited low-turnover osteoporosis
* lumbar spine or hip BMD T-score ≤ -2.5
* a written informed consent.

Exclusion Criteria:

* age less than 18 years
* generally accepted contraindications for the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in lumbar bone mineral density (BMD) | 0, 12 and 24 months
  The primary outcome measure is the change in lumbar BMD measured with dual-energy X-ray absorptiometry (DXA) during the 24 months treatment period.

SECONDARY OUTCOMES:
Change from baseline in whole body bone mineral density (DXA) | 0,12 and 24 months
Change from baseline in hip bone mineral density (DXA) | 0,12 and 24 months
Change from baseline in histomorphometry of bone biopsy samples | 0 and 24 months
  includes e.g following parameters: Bone volume (BV/TV, %); Osteoid volume (OV/BV, %); Trabecular thickness (Tb.Th, um); Osteoid surface (OS/BS, %); Osteoblast surface (Ob.S/BS, %); Eroded surface (ES/BS, %); Osteoclast surface (Oc.S/BS, %); Mineral apposition rate (MAR, um/day); Mineralizing surface (MS/BS, %)
Change from baseline in bone microarchitecture assessed by micro computed tomography of bone biopsy samples | 0 and 24 months
  includes e.g following parameters: bone volume (BV, mm3); relative bone volume (BV/TV, %); connectivity density, (Conn.D., 1/mm3); trabecular number (DT-Tb.N, 1/mm); trabecular thickness (DT-Tb.Th, mm)
Change from baseline in peripheral quantitative computed tomography (pQCT) measured cortical and trabecular volumetric bone mineral density of tibia and radius | 0,12 and 24 months
Number of vertebral fractures (spine X-ray) | 24 months
Change from baseline in serum procollagen type I N-terminal propeptide (PINP) | 0,3,6,12 and 24 months
Change from baseline in serum type I collagen C-telopeptides (CTX) | 0,3,6,12 and 24 months
Change from baseline in serum osteocalcin | 0,3,6,12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matti Välimäki, MD,PhD, Principal Investigator — Division of Endocrinology, Department of Medicine, Helsinki University Central Hospital
Locations (1):
- Department of Orthopaedics and Traumatology and Division of Endocrinology, Department of Medicine and Pediatric Endocrinology, Hospital for Children and Adolescents, Helsinki University Central Hospital, Helsinki, Finland